CLINICAL TRIAL: NCT04275401
Title: Study on Quantitative Evaluation of Muscle Tone Using Elastic Ultrasound
Brief Title: Quantitative Evaluation of Muscle Tone Using Elastic Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Mouwang Zhou, Professor, Peking University Third Hospital
Other Study IDs: M20191204
Record Dates: First submitted 2020-02-06; First posted 2020-02-19 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Muscle Tone Increased; Ultrasonography
MeSH Terms: conditions — Muscle Hypertonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients: patients with clinical presentions of change in muscle tone
- volunteers: healthy volunteers with normal muscle tone

SUMMARY:
The test subjects were selected from patients with clinical manifestations in muscle tone and healthy volunteers. Elbow flexor is the main target muscle. Fifty patients and 50 healthy subjects were given three assessment methods to measure muscle tension: modified Ashworth rating scale, elastic ultrasound technology and surface electromyography, and the data obtained by these three methods will be statistically analyzed and discussed.

ELIGIBILITY:
Inclusion Criteria:

* There are clinical manifestations of changes in muscle tension of the elbow flexor group;
* Subject's diagnosis is clear;
* The degree of joint mobility meets the method of muscle tension assessment.

Exclusion Criteria:

* Has serious diseases such as heart, lung, liver, kidney, etc., cardiac function grade is greater than Grade I (NYHA), has symptoms and signs or examination results such as respiratory failure;
* History of muscle disorders;
* Recent (within 6 months) history of external injury, fracture or surgery of the limb;
* Are using drugs that affect muscle tone;
* Severe osteoporosis;
* Acute phase of inflammation
* Acute limb thrombosis of the subject;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is expected to recruit 50 patients with clinical changes in flexion of the elbow flexor and 50 healthy subjects to participate in the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | through study completion, an average of 1 year
  Modified Ashworth Scale of the target muscles
shear wave elastography | through study completion, an average of 1 year
  use shear wave elastography to evaluate Young's modules of target muscles at each angle of the joint during the passive movement
surface electromyography | through study completion, an average of 1 year
  use surface electromyography to evaluate average EMG, integrated electromyogram and root mean square of the target muscles

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China